CLINICAL TRIAL: NCT01005095
Title: A One Year Prospective, Randomized, Double Blind Interventional Study to Assess Tolerability, Quality of Life and Immunomodulation With Interferon Beta Combined With Vitamin D in Patients With Relapsing Remitting Multiple Sclerosis
Brief Title: The Effects of Interferon Beta Combined With Vitamin D on Relapsing Remitting Multiple Sclerosis Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Interim analysis showed that the odds for proving primary hypothesis are low.
Sponsor: Carmel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RNFVD0209
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: MULTIPLE SCLEROSIS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High dose vitamin D (Experimental): 800 IU of Vitamin D3 by tablets plus a bottle of 75,000 IU vitamin D3 solution every 3 weeks
  Interventions: Dietary Supplement: Vitamin D3
- Low dose vitamin D (Active Comparator): 800 IU of vitamin D3 by tablets plus a 3 weekly placebo solution
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Patients will be treated daily with 800 IU of Vitamin D3 by tablets plus a bottle of 75,000 IU vitamin D3 solution every 3 weeks
  Arms: High dose vitamin D
Dietary Supplement: Vitamin D3 — Patients will receive 800 IU of vitamin D3 by tablets plus a 3 weekly placebo solution
  Arms: Low dose vitamin D

SUMMARY:
The investigators hypothesize that vitamin D supplementation may ameliorate interferon beta-induced flu-like symptoms, owing to reduced release and activity of the cytokines that are in correlation with this adverse event. Vitamin D supplementation may also positively affect injection site reactions due to its immunomodulatory effects. Vitamin D may also augment the therapeutic efficacy of interferon beta among multiple sclerosis (MS) patients. Vitamin D intake may influence melatonin levels of MS patients as they share the same nuclear receptor.

DETAILED DESCRIPTION:
Detailed Description of Study Evaluations

Adherence to treatment evaluation:

Patients will be asked to bring the empty packages of the IFN beta and Vitamin D that were used during the study.

Flu like symptoms and Injection site reactions evaluation:

Data regarding FLS and ISRs will be collected by means of a telephone interview every other week. The extent of FLS on the day of injection will be evaluated using a self-rating scale. A score from 0 (not at all) to 5 (very strong), will be given to each FLS component, i.e.: myalgia, chills, headache, malaise and fatigue, exacerbation of neurologic symptoms, sweating and difficulty to function compared to the time before injection. Patient will also record their oral temperature upon awakening as well as at their discretion. All patients will be provided with the same thermometer. Participants will be asked to report the frequency of Ibuprofen or Paracetamol use. and will be recommended not to exceed 800mg of Ibuprofen or 1000mg of Paracetamol per day, unless the symptoms are unbearable.

Patients will be inquired about the subjective degree of injection site pain for the first injections of every other week, by means of a 100 mm visual analogue scale (VAS scale). Patients will be seen at the clinic at 3 months intervals and in that visit the injection site will be inspected by the evaluating physician/ nurse and will be graded on a 0 to 3 scale: 0-none, 1- pain, itching or erythema, 2- swelling with inflammation and 3- ulceration and/or necrosis. Mode of application (manual or automatic injection) as well as needle size will be also recorded.

Patients will be instructed to refrain from reporting FLS and ISRs on the occasion of inter-current febrile illness or during and 4 weeks after corticosteroids treatment. In that case, patients will postpone the report by a week.

MS clinical parameters:

Patients will be clinically evaluated at enrollment and at 6 and 12 months for disease progression, by means of the EDSS score . The evaluating neurologist will be blinded to the patient's treatment.

Relapses, characterized by emergence of new symptoms or the worsening of existing ones for more than 24 hours in the absence of fever or infection ( McDonald et al., 2001) and severe enough to warrant corticosteroids treatment will be recorded.

Health related quality of life will be also evaluated at baseline and at the completion of the study, by means of a MS-specific validated questionnaire - FAMS (Functional Assessment of MS) (Miller A, 2006). (Attached)

Laboratory evaluation:

The following measurements will be obtained at the beginning of the study for the purpose of excluding patients with baseline impairment of mineral metabolism and at the end of the study to evaluate the resulting changes in mineral homeostasis consequent to vitamin D supplementation: blood levels of 25-OH- vitamin D, PTH, Magnesium, Calcium, Albumin, Creatinine, Urea, Phosphor, Alkaline phosphatase and 1-25- di-OH-D .

The following measurements will be assessed after 3, 6 and 12 months from study start for the purpose of 25-OH-D level monitoring and safety: Calcium, Phosphor, 25-OH-D , Albumin and creatinine. Laboratory evaluation required with IFN-beta safety will include: Complete blood count at baseline and after 3, 6, and 12 months from study start ; liver function tests at baseline and every 3 months, thyroid function tests at baseline, 6 months and by the end of the study or upon the emergence of symptoms suggestive of thyroid dysfunction.

Immunological markers:

Two venous blood samples will be drawn from a number of participants at Baseline and after 3 months of vitamin D supplementation . The first in the morning of IFN beta injection day and the second in the morning of the day after the injection. The percent rise after IFN beta injection of IL-6 and TRAIL will be assessed by commercial ELISA kits.

On visits baseline, 3 and 12 month, a venous blood portion will be stored at -80 oC within 30 min- 4 hour of blood withdrawal for MS related cytokines and proteins evaluation.

On visits baseline and 6 months another portion will be collected for immediately immune cell subset evaluation. PBMCs will isolated within 4 hour by Ficoll gradient centrifugation, stained with specific antibodies characterizing various immune cell subsets, and subset proportion determined by flow cytometry analysis.

Blood sampling will be postponed in case of a known condition that may possibly influence the expression of the studied cytokines. Namely, suspicion of a new or ongoing relapse within 30 days before or during the date of blood sampling; Clinical or paraclinical signs of acute infectious disease 48 hrs prior to blood sampling (leukocyte count > 10,000/mcl and /or CRP >2 mg/dl); Clinical signs of allergy within 7 days before participation; corticosteroids within 30 days before participation.

Melatonin:

Urine will be collected during 12-hour nighttime (20:00-08:00) at baseline, 3 months and by the end of the study. Levels of the melatonin metabolite (6-sulphatoxy-melatonin) will be assessed using a highly specific ELISA assay.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with a diagnosis of RRMS according to the McDonald criteria (2005)
* At least 18 years of age
* Patients are treated with IFN-beta for RRMS. The decision to treat with IFN beta will be independent from this study protocol.
* Patients will be either newly diagnosed, who are going to start IFN beta therapy for the first time or RRMS patients who suffer from FLS while being treated with IFN beta.
* Insufficient blood levels of 25-hydroxy-vitamin D (below 75nmol/l according to current definitions.
* EDSS score up to 7
* Willing and able to give informed consent

Exclusion Criteria:

* Patients having abnormalities of vitamin D related hormonal system other than low dietary intake or decreased sun exposure will be excluded. Namely, malabsorption [Celiac, Whipple, Inflammatory bowl disease, Intestinal bypass surgery, Short bowel syndrome, Cirrhosis, Nephrotic syndrome, Hyperthyroidism, Renal failure [creatinine clearance of less than 40 ml/min], Rickets, Hypoparathyroidism, Hypercalcemia at baseline, known malignancy, granulomatous disorders (Sarcoidosis, Tuberculosis, Silicosis) and Lymphomas.
* Patients who take medications that influence vitamin D metabolism, other than corticosteroids, will be also excluded. Namely, Orlistat, Anticonvulsants [Phenobarbital, Primidone, Phenytoin], Rifampin, Isoniazide, ketoconazole, 5FU and Leucovorin
* Patients with conditions with increased susceptibility to hypercalcemia will be excluded too: known arrhythmia or heart disease, treatment with Digitalis, or Hydrochlorothiazide.and those who suffer from nephrolithiasis.
* Other Central Nervous System disorders than RRMS
* Psychiatric disorders such as psychosis, bipolar disorder or substance abuse
* Pregnancy
* Contra-indication to treatment with IFN-beta

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Occurrence and severity of Interferon beta related Flu Like Symptoms and Injection Site Reactions. | One year

SECONDARY OUTCOMES:
Expanded Disability Status Scale (EDSS) progression | 1 year
Relapse rate | 1 year
Quality of life | 1 year
Change in serum levels of cytokines and proteins involved in MS pathogenesis | 12 months
Immune cells subsets | 6 months
Night time Urine levels of 6-sulphatoxy-melatonin | 1 year
Percent rise of IL6 and TRAIL levels following IFN-beta injection | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Miller, Prof, Principal Investigator — Multiple Sclerosis Center Carmel Medical Center
Locations (1):
- MS Clinic, Carmel Medical Center, Haifa, Israel, Israel

REFERENCES:
- [Derived] Golan D, Halhal B, Glass-Marmor L, Staun-Ram E, Rozenberg O, Lavi I, Dishon S, Barak M, Ish-Shalom S, Miller A. Vitamin D supplementation for patients with multiple sclerosis treated with interferon-beta: a randomized controlled trial assessing the effect on flu-like symptoms and immunomodulatory properties. BMC Neurol. 2013 Jun 14;13:60. doi: 10.1186/1471-2377-13-60. PMID 23767916